<u>Study identifiers:</u> DIAD Devic's Disease Auto 2008; NCT00787722 <u>Study title:</u> Hematopoietic Stem Cell Transplant in Devic's Disease

## Statistical Analysis

Time to progression and time to relapse were estimated via the Kaplan-Meier method and assessed via the log-rank test. Differences in outcome measures (EDSS, NRS, and SF-36) were compared by 2-tailed paired t test.